CLINICAL TRIAL: NCT01668615
Title: Efficacy of Immunomudulatory Therapy With All-trans Retinoid Acid for Adults With Chronic Immune Thrombocytopenia
Acronym: ITP
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Suzhou Medical College (Other)
Responsible Party: Principal Investigator, Zhaoyue Wang, Jiangsu Institute of hematology, First Affiliated Hospital of Suzhou Medical College
Other Study IDs: jsxys-123
Record Dates: First submitted 2012-07-30; First posted 2012-08-20 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: idiopathicthrombocytopenic purpura; all-trans retinoic acid; regulory T cells
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Tretinoin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: all-trans-retinoid acid — 10 mg three times a day oral administration for 4 months
  Other Names: Tretinoin

SUMMARY:
The purpose of this study is to determine whether All-trans retinoic acid (ATRA) are effective in the treatment of refractory idiopathic thrombocytopenic purpura (RITP).

DETAILED DESCRIPTION:
Idiopathic thrombocytopenic purpura(ITP), an acquired immune disease is characterized by impaired generation of autoantibody-specific platelet. At least 30% adult patients turn into refractory ITP. The pathogenesis of ITP remains to be elucidated. Now ,CD4+ helper cells have been classified as belong to T-helper 1(TH1), T-helper 2(TH2), T-helper17and Regulory T cell(Tregs). All-trans retinoic acid(ATRA) mainly applied in skin disease and acute promyelocytic leukemia. Recently, ATRA is also a immunomodulator which can induce differentiation, proliferation, apoptosis of cells, and immunomudulatory. In the international, the investigators first treat RITP with ATRA. To investigate the therapeutic effects of ATRA on RITP, and using new index in the cells, cytokines and molecular biology of three in-depth study of its mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of refratory idiopathic thrombocytopenic purpura
* Hormone and immune suppression, splenectomy is invalid

Exclusion Criteria:

* Other autoimmune diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 35 patients of RITP who do not response to prednisone,immunosuppressive agents and/or splenectomy were observed in our study .
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: zhaoyue wang, doctor, Study Director
Locations (1):
- Jiangsu Institute of Hematology, Suzhou, Jiangsu, China